CLINICAL TRIAL: NCT02340572
Title: A First-in-Human, Randomized, Dose-Escalation, Double-Blind, Placebo-Controlled Single Ascending Dose Study to Establish Safety, Lack of Immunogenicity, Tolerability, Pharmacokinetic Parameters, Target Engagement and Pharmacodynamic Effects
Brief Title: First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PRS-080
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pieris Pharmaceuticals GmbH (Industry)
Collaborators: Nuvisan Pharma Services (Unknown); FGK Clinical Research GmbH (Industry); EUROCALIN Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: PCS_01_12
Record Dates: First submitted 2014-12-18; First posted 2015-01-16 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRS-080#022-DP (Experimental): hepcidin antagonist, single administration, ascending doses
  Interventions: Drug: PRS-080#022-DP
- PRS-080-Placebo#001 (Placebo Comparator): Comparotor treatment, single administration
  Interventions: Drug: PRS-080-Placebo#001

INTERVENTIONS:
Drug: PRS-080#022-DP — hepcidin antagonist
  Other Names: PRS-080
  Arms: PRS-080#022-DP
Drug: PRS-080-Placebo#001 — Placebo treatment
  Other Names: Placebo
  Arms: PRS-080-Placebo#001

SUMMARY:
Anticalins® are engineered human proteins that are able to bind specific target molecules. The Anticalin PRS-080#022-DP to be investigated in this study is directed against hepcidin and is intended for treatment of anemia of chronic disease. This phase I First-in-Human study shall investigate safety and pharmacokinetics in healthy human volunteers.

DETAILED DESCRIPTION:
First-in-Human (FIH), randomized, dose-escalation, double-blind, placebo-controlled single dose in healthy volunteers.

The single rising dose study will enroll 8 subjects per cohort (6 verum, 2 placebo), up to a maximum tolerated dose, defined by stopping rules. 6 dose levels are anticipated. Study drug will be administered as i.v. infusion on Day 1. The decision to escalate the dose by the dose escalation committee (DEC) will be based on an interim analysis of clinical safety and safety laboratory data.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Caucasian males: based on a screening examination including medical history, physical examination, 12-lead ECG, vital signs and clinical laboratory profiles, age 18-50 years
2. Subjects should have a body mass index of 18-30 kg/m2 and should weigh 60-90 kg
3. Subjects must be using two acceptable methods for contraception (e.g. spermicide and condom) during the study and refrain from fathering a child in the 3 months following the last dosing.
4. Willing to comply with the requirements of the study protocol and signing the informed consent sheet.

Exclusion Criteria:

1. Any uncontrolled or active major systemic disease
2. History or presence of malignancy
3. Definite or suspected history of drug allergy
4. Active acute or chronic infection, including, but not limited to: upper airway infection, urinary tract infection, and skin infection
5. Use of any investigational drug within 30 days, or 5 half-lives, whichever is longer, prior to the planned first drug administration.
6. Use of prescription medication within 14 days prior to the planned first drug administration and throughout the study (with the exception of medications given to treat an adverse event and use of non-prescription or over-the-counter medications within 7 days prior to the planned first drug administration and throughout the study (including vitamins, herbal supplements, or remedies
7. Smoking greater than 20 cigarettes per week
8. History of alcohol or substance abuse within the past 6 months prior to the planned first drug administration
9. History of increased bleeding risk
10. Clinically relevant abnormalities found in physical examination, vital signs measurements, laboratory safety tests or ECG
11. Blood donation within the last 60 days prior to the planned first drug administration
12. Positive results on hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV1/2) antibodies screening
13. Iron overload or disturbance in utilization of iron (defined as ferritin > 300.0 ng/mL and < 10.0 ng/mL)
14. i.v. iron treatment or blood transfusion within last 90 days prior to the planned first drug administration or during trial
15. ESA (e.g. Erythropoietin) treatment within the last year
16. Surgery or trauma with significant blood loss within 2 months before the planned first drug administration
17. Not able to abstain from consumption of food or beverages known to influence dietary iron absorption

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 28 days
  Composite measure including signs and symptoms, local reactions, changes from baseline heart rate and blood pressure, ECG, body temperature, respiratory rate, clinical chemistry and hematology, coagulation and urinalysis over a 28 day period

SECONDARY OUTCOMES:
Pharmacokinetics of PRS-080#22-DP following administration of single doses | 14 time points up to 11 days
  Area under the plasma concentration versus time curve (AUC) of PRS-080#22-DP in blood
Assessment of anti-drug antibodies in blood following single administration | up to 28 days
  Analysis of antibodies against PRS-080#22-DP at day 28 compared to baseline
Effect of PRS-080#22-DP on hepcidin concentrations in blood | 15 time points up to 28 days
  Changes in hepcidin concentration compared to baseline
Effect of PRS-080#22-DP on total iron | up to 28 days
  Changes in total iron concentration in blood compared to baseline
Effect of PRS-080#22-DP on transferrin saturation | up to 28 days
  Changes in transferrin saturation in blood compared to baseline
Effect of PRS-080#22-DP on ferritin | up to 28 days
  Changes to ferritin concentration in blood compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Moebius, PhD, Study Director — Pieris Pharmaceuticals GmbH
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany